CLINICAL TRIAL: NCT02348411
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound for Bilateral Anterior Capsulotomy in the Treatment of Medication-Refractory MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2014-0073
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Diorder
Keywords: Medication-refractory
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate Treatment group (Experimental)
  Interventions: Device: ExAblate

INTERVENTIONS:
Device: ExAblate
  Other Names: Treatment with the ExAblate Transcranial MRgFUS System

SUMMARY:
The purpose of this study is to evaluate the safety and initial effectiveness of MRI-guided focused ultrasound thermal ablation of a designated area in the brain of patients suffering from medication-refractory MDD, using the ExAblate transcranial system.

The ExAblate system is a medical device that involves a focused ultrasound system and an MRI scanner. ExAblate delivers a pulse of focused ultrasound energy, or sonication, to the targeted tissue. For MDD Patients: one or more thermal lesion will be created on Bilateral Anterior Limb of internal Capsule.

The treatment begins with a series of standard diagnostic MR images to identify the location and shape of target to be treated. The ExAblate computer uses the physician's designation of the target volume to plan the best way to cover the target volume with small spots called "sonications". These treatment spots are cylinder shaped. Their size depends on sonication power and duration. During the treatment, a specific MR scan, which can be processed to identify changes in tissue temperature, provides a thermal map of the treatment volume to confirm the therapeutic effect. The thermal map is used to monitor the treatment in progress, and confirm that the ablation is proceeding according to plan, thus closing the therapy loop.

The ExAblate transcranial operates a helmet-shaped transducer (currently utilizing 1000-element phased array transducer) positioned above the subject head. The ExAblate transcranial system also includes means to immobilize the subject head, cool the interface water, and software for CT analysis and phase correction computation.

After informed consent and screening, eligible subjects will proceed to the treatment. All subjects will be followed at Day 1, 7 days, 1 month , and 6 months . At follow up visits, patients will be evaluated for general health, neurological changes (including MMSE exam),and efficacy measurements as well as for device/procedure related adverse events that may have occurred during the follow-up period. Six (6) month follow up visit will also include Full Battery Cognitive/Neurological Testing

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 20 and 65 years, inclusive
* Diagnosed with nonpsychotic major depressive disorder, single or recurrent episode by DSM-IV-TR Diagnosis of Diagnostic and Statistical Manual of Mental Disorder fourth edition(DSM-IV) MDD as confirmed from clinical history and examination by psychiatrist.
* Subjects who are able and willing to give consent and able to attend all study visits
* Proof of Refractoriness

In current episode:

* Depression refractory to adequate trials of medication (Persistence of the major depressive episode to a minimum of 3 adequate depression treatments from at least 3 different treatment categories - SSRIs, TCAs, other antidepressants, lithium addition, irreversible MAO inhibitor, etc.)
* Documented resistance to ECT (at least 6 sessions or <6 treatments if there is clear evidence of inability to tolerate more, or refused, or withdrew consent after ECT was recommended.

  - Proof of chronicity
* More than 5 years after first episode of MDD
* current episode of ≥24-mo duration &/or recurrent illness with at least a total of 4 lifetime episodes (including current episode ≥12 mos)

  - Proof of Severity
* HAMD-17 score≥20
* Global Assessment of Function Score<50

  * Designated Ablation Targets can be target by the ExAblate device. Designated Ablation Targets must be apparent on MRI such that targeting can be performed with direct visualization
  * Able to communicate sensations during the ExAblate MRgFUS treatment
  * Depression medication regimen is stable for at least 30 days before enrollment

Exclusion Criteria:

* Subjects with current or previous diagnosis of following psychotic or bipolar disorders:
* Subjects has primary or serious(requiring additional treatment) comorbid obsessive compulsive disorder, posttraumatic stress disorder, panic disorder, bulimia, or anorexia in the last year by DSM-IV
* Patients exhibiting any behavior(s) consistent with ethanol or substance abuse(aside nicotine) as defined by the criteria outlined in the DSM-IV occurring within a 12 months period
* Active suicidal ideation with plan or intent for self harm and made suicide attempt within the past 12 months
* Patient meets criteria for personality disorder in the last 12 months by DSM-IV
* Patients with unstable cardiac status including:

  * Unstable angina pectoris on medication
  * Patients with documented myocardial infarction within six months of protocol entry
  * Congestive heart failure requiring medication (other than diuretic)
  * Patients on anti-arrhythmic drugs
* Severe hypertension (diastolic BP > 100 on medication)
* Severely impaired renal function (estimated glomerular filtration rate < 45ml/min/1.73 m2) or receiving dialysis
* Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent(e.g. Gadolinium or Magnevist) including advanced kidney disease
* History of abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
* Active or suspected acute or chronic uncontrolled infection
* History of intracranial hemorrhage
* Cerebrovascular disease (multiple CVA or CVA within 6 months)
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
* Symptoms and signs of increased intracranial pressue (e.g. headache, nausea, vomiting, lethargy, and papilledema)
* Are participating or have participated in another clinical trial in the last 30 days
* Unable to communicate with the investigator and staff.
* Presence of any other neurodegenerative disease like Parkinson-plus syndromes suspected on neurological examination. These included:

  * Multisystem atrophy
  * Progressive supranuclear palsy
  * Dementia with Lewy bodies
  * Alzheimer's disease
* Anyone suspected to have the diagnosis of MDD. This includes: psychotic depression, bipolar I or II disorder, mental disorder due to organic factors.
* Presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
* History of immunocompromise, including patient who is HIV positive
* Known life-threatening systemic disease
* Patients with a history of seizures within the past year
* For the purpose of this study, we consider a significant mood disorder to include any patient who has:

  * received transcranial magnetic stimulation
  * received electroconvulsive therapy
* Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter, PT > 14, PTT > 36 or INR > 1.3) or a documented coagulopathy
* Patients with any types of brain tumors, including metastases.
* Any illness that in the investigator's opinion preclude participation in this study.
* Pregnancy or lactation.
* Legal incapacity or limited legal capacity.
* Patients who have had deep brain stimulation or a prior stereotactic ablation of the Designated Ablation Target.
* Prior intracranial surgery
* Calcifications in the sonication pathway that cannot be avoided by tailoring the treatment plan
* More than 30% of the scalp in the sonication pathway is covered by scars, scalp disorders (e.g., eczema) or atrophy of the scalp
* Clips or other metallic implanted objects in the sonication pathway, except shunts.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
To assess Hamilton Depression Rating Scale-17 | 6 months

SECONDARY OUTCOMES:
To assess adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim M, Kim CH, Jung HH, Kim SJ, Chang JW. Treatment of Major Depressive Disorder via Magnetic Resonance-Guided Focused Ultrasound Surgery. Biol Psychiatry. 2018 Jan 1;83(1):e17-e18. doi: 10.1016/j.biopsych.2017.05.008. Epub 2017 May 12. No abstract available. PMID 28601192